CLINICAL TRIAL: NCT04722484
Title: Investigation of Pharmacokinetics, Safety, Tolerability and Pharmacodynamic Effects of BAY1021189 in Male and Female Subjects With Renal Impairment and in Age-, Gender-, and Weight-matched Healthy Subjects Following a Single Oral Dose of 2.5 mg BAY1021189 in a Single-center, Non Randomized, Non-controlled, Non-blinded, Observational Study With Group Stratification
Brief Title: A Trial to Learn How Safe Vericiguat (BAY1021189) is and the Way the Body Absorbs, Distributes and Gets Rid of Vericiguat in Participants With Kidney Disease and in Age-, Weight- and Gender-matched Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15813; 2013-004762-34 (EudraCT Number)
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — vericiguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Patients with normal creatine clearance (CLCR) (Experimental): Subjects with renal impairment according to their medical history and estimated glomerular filtration rate (eGFR) at screening but had normal creatinine clearance at the pre-profile day (-01day)
  Interventions: Drug: Vericiguat (BAY1021189)
- Normal renal function (Healthy subjects) (Experimental): Subjects with creatinine clearance at pre-profile day >80 ml/min
  Interventions: Drug: Vericiguat (BAY1021189)
- Mildly impaired renal function (Experimental): Subjects with creatinine clearance at pre-profile day in the range of 50-80 ml/min
  Interventions: Drug: Vericiguat (BAY1021189)
- Moderately impaired renal function (Experimental): Subjects with creatinine clearance at pre-profile day in the range of 30-<50 ml/min
  Interventions: Drug: Vericiguat (BAY1021189)
- Severely impaired renal function (Experimental): Subjects with creatinine clearance at pre-profile day <30 ml/min
  Interventions: Drug: Vericiguat (BAY1021189)

INTERVENTIONS:
Drug: Vericiguat (BAY1021189) — Oral single dose of 2.5 mg (2 x 1.25 mg immediate release tablet)

SUMMARY:
Vericiguat (BAY1021189) is under development to treat heart failure, a condition in in which the heart has trouble pumping blood through the body. Renal impairment which co-occurs in patients with heart failure is a common condition in which the kidneys are not filtering the blood as well as they should.

The goal of the study was to learn more about the safety of vericiguat (BAY1021189), how it was tolerated and the way the body absorbed, distributed and excreted the study dug given as a single oral dose of 2.5 mg tablet in participants with renal impairment and healthy participants matched for age-, gender-, and weight.

The participants stayed at the trial site for about 6 days. During this time, the doctors took blood and urine samples and checked the participants' health. About 7-14 days after the participants took vericiguat (BAY1021189), the researchers checked the participants' health again and asked about any medical problems they had.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Aged between 18 and 79 years (inclusive) with body mass index 18 to 34 kg/m^2 (both inclusive)
* Women without childbearing potential; women of childbearing potential only if the pregnancy test was negative and a combination of condoms with a safe and highly effective contraception method was granted

For subjects with renal impairment:

* With an estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73m^2 determined from a serum creatinine control 2-14 days prior to dosing
* Stable renal disease, i.e. a serum creatinine value determined at least 3 months before the pre-study visit should not vary by more than 25% from the serum creatinine value determined at the pre-study visit

For healthy subjects:

* eGFR ≥ 90 mL/min/1.73m^2 determined from serum creatinine 2-14 days prior to dosing
* Healthy subjects with age-, weight- and gender- matched to renal impaired subjects

Exclusion Criteria:

For all subjects:

* Febrile illness within 1 week before the start of the study
* History of severe allergies, non-allergic drug reactions, or multiple drug allergies
* Hypersensitivity to the investigational drug, the control agent and/ or to inactive constituents
* Regular daily consumption of more than 1/2 liter of usual beer or the equivalent quantity of approximately 20 g of alcohol in another form or more than 1 liter of xanthine-containing beverages or more than 10 cigarettes
* Positive testing in the drug screening
* Positive results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), human immune deficiency virus antibodies (anti-HIV 1+2)
* Donation of more than 100 mL of blood in the preceding 4 weeks or 500 mL in the preceding 3 months
* Relevant deviation from the normal range in clinical chemistry, hematology, coagulation or urinalysis as judged by the investigator For subjects with renal impairment
* Acute renal failure
* Acute nephritis
* Any organ transplant in the past 5 years
* Severe cerebrovascular or cardiac disorders, e.g. myocardial infarction less than 6 months prior to dosing, congestive heart failure of New York Heart Association grade III or IV, severe arrhythmia requiring anti-arrhythmic treatment
* Percutaneous transluminal coronary angioplasty or coronary artery bypass graft less than 6 months prior to dosing
* Diagnosed malignancy within the past 5 years
* Failure of any other major organ system other than the kidney
* Concomitant use of any medication except medications necessary for the treatment of diseases
* Diastolic BP >100 mmHg and/or systolic BP >180 mmHg
* Heart rate below 50 beats/min or above 100 beats/min at screening visit
* Significant uncorrected rhythm or conduction disturbances For healthy subjects
* Subjects with conspicuous findings in medical history or pre-study examination
* A history of relevant diseases of vital organs, of the central nervous system or other organs
* Excluded therapies (e.g. physiotherapy, acupuncture, etc.) from 1 week before admission to the ward (-01d)
* Use of medication within the 2 weeks preceding the study which could interfere with the investigational product
* Systolic BP below 100 mmHg or above 145 mmHg and Diastolic BP below 55 mmHg or above 95 mmHg
* Heart rate below 50 beats/min or above 100 beats/min
* Clinically relevant findings in the electrocardiogram (ECG)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-06-12 (Actual); Primary Completion 2015-01-22 (Actual); Study Completion 2015-01-22 (Actual)

PRIMARY OUTCOMES:
AUC of vericiguat | Up to 96 hours
  Area under the concentration vs. time curve from zero to infinity after single dose administration
Cmax of vericiguat | Up to 96 hours
  Maximum observed drug concentration in measured matrix after single dose administration
AUC of vericiguat's metabolite M-1 | Up to 96 hours
  Area under the concentration vs. time curve from zero to infinity after single dose administration
Cmax of vericiguat's metabolite M-1 | Up to 96 hours
  Maximum observed drug concentration in measured matrix after single dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Kiel, Schleswig-Holstein, Germany

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/